CLINICAL TRIAL: NCT03891199
Title: A Two Year Multicenter Study of Robotic-Arm Assisted THA: Acetabular Cup Placement Accuracy and Clinical Outcomes
Brief Title: Two Year Study With Robotic-Arm Assisted Hip Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Stryker Nordic (Industry); West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Matthew Dietz, MD, Associate Professor, Chair, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1808218345
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Surgery; Hip Osteoarthritis
Keywords: clinical trial; randomization; hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Traditional THA.
- Intervention (Active Comparator): Robotic-arm assisted THA.
  Interventions: Procedure: Robotic-Arm Assisted THA

INTERVENTIONS:
Procedure: Robotic-Arm Assisted THA — The study will examine the acetabular cup placement of THA patients and compare results for patients who undergo THA with robotic-arm assistance with those who undergo traditional THA.
  Arms: Intervention

SUMMARY:
This study will involve a quantitative assessment of prospectively collected computed tomography, radiographic and patient outcomes data from multiple centers. Specifically looking at acetabular cup placement during Total Hip Arthroplasty by either traditional or robotic-arm assisted placement.

DETAILED DESCRIPTION:
The incidence of dislocation following total hip arthroplasty (THA) has been reported to be from 1% to as much as 3.2%. The demand for THA is expected to increase. Post- dislocation solutions include closed reduction, open reduction, THA revision, and constrained cup, conversion to hemiarthroplasty, allograft or girdlestone resection. These solutions are often costly, painful and can involve substantial additional risks and complications. Acetabular cup placement is an important factor in the stability of the THA. Cup malpositioning has been associated with bearing surface ware and dislocation. For most patients, acceptable angles for abduction are 40° abduction (±10°) and 20° (±5°) version. However, malpositioning continues to occur resulting in cup angles outside acceptable ranges and leaving patients with an increased risk of dislocation.

This objective of this study is to examine the acetabular cup placement of THA patients and compare results for patients who undergo THA with robotic-arm assistance with those who undergo traditional THA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring primary total hip arthroplasty
2. Patients willing and able to comply with follow-up requirements
3. Patients willing to sign an Institutional Review Board approved informed consent form.

Exclusion Criteria:

1. Patients with Body Mass Index >45
2. Patients who are <18 years of age
3. Patients with an active infection or suspected latent infection in or about the hip joint
4. Bone stock that is inadequate for support or fixation of the prosthesis
5. Previous major hip surgery excluding hip arthroscopy
6. Total hip arthroplasty using cement fixation or resurfacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Dietz, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Medicine, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All patient outcomes data will be entered by the on-site research assistant into the REDCap study site created and managed at the Principal Investigators institution by the primary research coordinator. The REDCap site will house the study data and provide a means for the remote site research assistant to enter patient demographics, medical history, surgical details and outcome results. Medical history, demographic, and surgical details.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The individual participant data (IPD) will be available from the beginning of enrollment until the manuscript is submitted and accepted
Access Criteria: the study will utilize a digital imaging analysis program called the Martell Hip Analysis Suite (HAS, Chicago, IL) as well as Computed Tomography (CT) scans. Patient reported outcomes (HOOS, PROMIS10, Hip stability and return to function) will also be collected at specified intervals. Using CT Scans and HAS analysis allows for a complete description of cup placement, and better accounts for factors such as pelvic rotation and/or tilt, otherwise not accounted for in radiographic analysis.

REFERENCES:
- [Background] Banerjee S, Cherian JJ, Elmallah RK, Pierce TP, Jauregui JJ, Mont MA. Robot-assisted total hip arthroplasty. Expert Rev Med Devices. 2016;13(1):47-56. doi: 10.1586/17434440.2016.1124018. Epub 2015 Dec 21. PMID 26592900
- [Background] Elson L, Dounchis J, Illgen R, Marchand RC, Padgett DE, Bragdon CR, Malchau H. Precision of acetabular cup placement in robotic integrated total hip arthroplasty. Hip Int. 2015 Nov-Dec;25(6):531-6. doi: 10.5301/hipint.5000289. Epub 2015 Sep 10. PMID 26391264
- [Background] Kanawade V, Dorr LD, Banks SA, Zhang Z, Wan Z. Precision of robotic guided instrumentation for acetabular component positioning. J Arthroplasty. 2015 Mar;30(3):392-7. doi: 10.1016/j.arth.2014.10.021. Epub 2014 Oct 22. PMID 25453633
- [Background] Werner SD, Stonestreet M, Jacofsky DJ. Makoplasty and the accuracy and efficacy of robotic-assisted arthroplasty. Surg Technol Int. 2014 Mar;24:302-6. PMID 24574012
- [Background] Tarwala R, Dorr LD. Robotic assisted total hip arthroplasty using the MAKO platform. Curr Rev Musculoskelet Med. 2011 Sep;4(3):151-6. doi: 10.1007/s12178-011-9086-7. PMID 21728013
- [Background] Callanan MC, Jarrett B, Bragdon CR, Zurakowski D, Rubash HE, Freiberg AA, Malchau H. The John Charnley Award: risk factors for cup malpositioning: quality improvement through a joint registry at a tertiary hospital. Clin Orthop Relat Res. 2011 Feb;469(2):319-29. doi: 10.1007/s11999-010-1487-1. PMID 20717858
- [Background] Woo RY, Morrey BF. Dislocations after total hip arthroplasty. J Bone Joint Surg Am. 1982 Dec;64(9):1295-306. PMID 7142237
- [Background] Lewinnek GE, Lewis JL, Tarr R, Compere CL, Zimmerman JR. Dislocations after total hip-replacement arthroplasties. J Bone Joint Surg Am. 1978 Mar;60(2):217-20. PMID 641088
- [Background] Domb BG, El Bitar YF, Sadik AY, Stake CE, Botser IB. Comparison of robotic-assisted and conventional acetabular cup placement in THA: a matched-pair controlled study. Clin Orthop Relat Res. 2014 Jan;472(1):329-36. doi: 10.1007/s11999-013-3253-7. Epub 2013 Aug 29. PMID 23990446
- [Background] Banerjee S, Cherian JJ, Elmallah RK, Jauregui JJ, Pierce TP, Mont MA. Robotic-assisted knee arthroplasty. Expert Rev Med Devices. 2015;12(6):727-35. doi: 10.1586/17434440.2015.1086264. Epub 2015 Sep 12. PMID 26365088
- [Background] Roche M. Robotic-assisted unicompartmental knee arthroplasty: the MAKO experience. Orthop Clin North Am. 2015 Jan;46(1):125-31. doi: 10.1016/j.ocl.2014.09.008. PMID 25435041
- [Background] Soong M, Rubash HE, Macaulay W. Dislocation after total hip arthroplasty. J Am Acad Orthop Surg. 2004 Sep-Oct;12(5):314-21. doi: 10.5435/00124635-200409000-00006. PMID 15469226
- [Background] Pellicci PM, Bostrom M, Poss R. Posterior approach to total hip replacement using enhanced posterior soft tissue repair. Clin Orthop Relat Res. 1998 Oct;(355):224-8. doi: 10.1097/00003086-199810000-00023. PMID 9917607
- [Background] Ghelman B, Kepler CK, Lyman S, Della Valle AG. CT outperforms radiography for determination of acetabular cup version after THA. Clin Orthop Relat Res. 2009 Sep;467(9):2362-70. doi: 10.1007/s11999-009-0774-1. Epub 2009 Mar 10. PMID 19277802
- [Background] Redmond JM, Gupta A, Hammarstedt JE, Petrakos A, Stake CE, Domb BG. Accuracy of Component Placement in Robotic-Assisted Total Hip Arthroplasty. Orthopedics. 2016 May 1;39(3):193-9. doi: 10.3928/01477447-20160404-06. Epub 2016 Apr 12. PMID 27064781
- [Background] El Bitar YF, Stone JC, Jackson TJ, Lindner D, Stake CE, Domb BG. Leg-Length Discrepancy After Total Hip Arthroplasty: Comparison of Robot-Assisted Posterior, Fluoroscopy-Guided Anterior, and Conventional Posterior Approaches. Am J Orthop (Belle Mead NJ). 2015 Jun;44(6):265-9. PMID 26046996
- [Background] Gupta A, Redmond JM, Hammarstedt JE, Petrakos AE, Vemula SP, Domb BG. Does Robotic-Assisted Computer Navigation Affect Acetabular Cup Positioning in Total Hip Arthroplasty in the Obese Patient? A Comparison Study. J Arthroplasty. 2015 Dec;30(12):2204-7. doi: 10.1016/j.arth.2015.06.062. Epub 2015 Jul 2. PMID 26253480
- [Background] Bukowski BR, Anderson P, Khlopas A, Chughtai M, Mont MA, Illgen RL 2nd. Improved Functional Outcomes with Robotic Compared with Manual Total Hip Arthroplasty. Surg Technol Int. 2016 Oct 26;29:303-308. PMID 27728953
- [Background] Kamara E, Robinson J, Bas MA, Rodriguez JA, Hepinstall MS. Adoption of Robotic vs Fluoroscopic Guidance in Total Hip Arthroplasty: Is Acetabular Positioning Improved in the Learning Curve? J Arthroplasty. 2017 Jan;32(1):125-130. doi: 10.1016/j.arth.2016.06.039. Epub 2016 Jun 29. PMID 27499519

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 20 | 20
Completed | 20 | 17
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 10 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 17 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Acetabular Cup Placement Manually vs. Robotic-arm Assisted - Version.
Description: Accuracy of cup placement will be measured by absolute value of degrees from target version (40 degrees). Using CT (Computed Tomography) Scans, analysis and radiographs will allow for a complete description of cup placement, and better accounts for factors such as pelvic rotation and/or tilt, otherwise not accounted for in radiographic analysis alone.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees error in anteversion
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 17
degrees error in anteversion | 5.95 (2.78) | 4.26 (3.19)

2. Primary Outcome: Change in Patient Reported "Hip Dysfunction and Osteoarthritis Outcome Score" (HOOS) Survey Over 1 Year Period.
Description: The hip disability and osteoarthritis outcome score (HOOS) is a questionnaire intended to be used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process . To interpret the score, the outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms. To calculate the total HOOS score the subscales need to be summed up.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 17
score on a scale
  HOOS Pain Improvement | 39.54 (9.98) | 47.92 (6.34)
  HOOS ADL (activities of daily living) | 41.31 (9.98) | 48.40 (4.59)
  HOOS Symptoms | 32.27 (10.65) | 59.17 (4.99)
  HOOS QOL (quality of life) | 43.75 (11.46) | 53.13 (9.05)
  HOOS Sports/recreation | 31.82 (12.93) | 58.85 (6.63)

3. Primary Outcome: Change in "Patient-Reported Outcomes Measurement Information System" (PROMIS) Survey Over a 1 Year Period.
Description: The PROMIS Global-10 is a global health quality of life patient reported outcome tool. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS). It measures symptoms, functioning, and healthcare quality of life for a wide variety of conditions. The PROMIS Global-10 consists of 10 questions assessing physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. 7 questions inquire about health in "general" and 3 questions assess emotional problems, fatigue and pain in the last 7 days.
  PROMIS 10 Global Physical Health- Scale range (0-20) and what the low number means vs the high number (ex 0 equals worse physical health and 20 equals the best physical health). PROMIS 10 Global Mental Health- Scale range (0-20) and what the low number means vs the high number (ex 0 equals worse mental health and 20 equals the best mental health)
Time Frame: 1year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 17
score on a scale
  PROMIS 10 Global Physical Health | 10.11 (3.01) | 11.37 (2.72)
  PROMIS 10 Global Mental Health | 3.92 (3.38) | 2.88 (1.73)

4. Primary Outcome: Accuracy of Acetabular Cup Placement Manually vs. Robotic-arm Assisted - Inclination.
Description: Accuracy of cup placement will be measured by absolute value of degrees from target inclination (20 degrees). Using CT (Computed Tomography) Scans, analysis and radiographs will allow for a complete description of cup placement, and better accounts for factors such as pelvic rotation and/or tilt, otherwise not accounted for in radiographic analysis alone.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees error in inclination
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 17
degrees error in inclination | 4.73 (3.58) | 2.93 (2.42)

5. Primary Outcome: Adherence to Lewinnek Safe Zone
Description: 5-25 degrees of anteversion; 30-50 degrees of inclination.
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 20 | 17
Participants
  version in the Lewinnek safe zone | 14 | 16
  inclination in the Lewinnek safe zone | 17 | 17

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=20) | Intervention (N=20)
Prosthetic Joint Infection (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03891199/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03891199/ICF_001.pdf